CLINICAL TRIAL: NCT01942850
Title: APPLICABILITY OF THE INTERNATIONAL ATAXIA RATING SCALE (ICARS) IN YOUNGER PATIENTS AND DEVELOPMENT OF GLOBAL RATING INSTRUMENTS FOR PATIENTS WITH ATAXIA TELANGIECTASIA (AT)
Brief Title: International Ataxia Rating Scale in Younger Patients
Status: Completed | Type: Observational
Sponsor: Quince Therapeutics S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: ICARS-CGI-Ery01-2013
Record Dates: First submitted 2013-09-06; First posted 2013-09-16 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Ataxia Telangiectasia
MeSH Terms: conditions — Ataxia Telangiectasia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No Treatment: Collect pilot data on the performance of the ICARS in patients younger than 10 years of age, as well as to introduce definitions for the various clinically defined stages of AT, and attempt to develop descriptors of change that could help in the assessment of patients longitudinally.

SUMMARY:
The project will collect information on the mapping of clinical ratings on a number of scales that are used in the assessment of patients with ataxias.

ELIGIBILITY:
Inclusion criteria

1. Patients aged 6-18 years with diagnosed with ataxia, preferably AT will be included. The diagnosis of AT will be made based on the criteria: typical clinical picture plus one of the following: 1. a proven mutation in the ATM gene 2. Deficient ATM protein proven by Western blotting 3. Elevated α-fetoprotein, cerebellar atrophy on MRI and immune deficiency/ chromosomal breakage/ T- cell lymphoreticular malignancy.
2. Children aged 6-18 years with suspected AT (fulfilling partially the above criteria will be included)
3. Children aged 6-18 years with AT like disease, with or without proven mutation in the MRE11 gene will be included
4. Children aged 6-18 years of age with ataxia of other known or unknown etiologies might be included, but their total number should not exceed 20% of the cohort in each site

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Known patients with ataxia/ataxia telangiectasia
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Correlation Analysis | single visit
  The primary outcome is validity of ICARS in children younger than 10 years of age (by comparing the mean scores and subscores between children aged 6-10 years of age to those aged 10-18 years of age).

CONTACTS AND LOCATIONS:
Overall Officials: Luca Benatti, MD, Study Director — Quince Therapeutics S.p.A.
Locations (5):
- Carol Morsani USF Health Center, Tampa, Florida, United States
- Jaslok Hospital, Mumbai, India
- Edmond and Lilly Safra Childrens Hospital Pediatric Unit, Tel Litwinsky, Israel
- Italy (2):
  - Università La Sapienza, Roma, Italy
  - A.O Spedalli Civilli Brescia, Brescia